CLINICAL TRIAL: NCT04010318
Title: The Sensitivity of Goal Plethysmography Variability Index (PVI) Directed Pre-anesthesia Intravenous Fluid Infusion in the Prevention of Spinal Anesthesia Induced Hypotension in Elective Caesarian Section: Prospective Observational Study
Brief Title: Plethysmographic Variability Index in Post Spinal Anesthesia Hypotension in Cesarean Section
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Collaborators: Tamer Mohamed Naguib (Unknown); Amr Ahmed Magdy (Unknown)
Responsible Party: Principal Investigator, Sameh Abdelkhalik Ahmed Ismaiel, Dr, Tanta University
Other Study IDs: 33109/05/19
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Complication of Anaesthesia During Labour and Delivery
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Corrected group: The patients in which the PVI will corrected by fluid to level below 15
  Interventions: Procedure: Spinal Anesthesia
- Uncorrected group: Patients in which intravenous fluid administration didn't result any change in PVI or changed but still higher than 15
  Interventions: Procedure: Spinal Anesthesia

INTERVENTIONS:
Procedure: Spinal Anesthesia — The patients will receive spinal block at lumbar 3-4 space with hyperbaric bupivacaine 8 mg plus 25 mic fentanyl. After giving anesthesia and positioning for surgery with a left lateral tilt of 15 degrees, supplemental oxygen at rate of 4 liter/minute is applied.

SUMMARY:
* Full term pregnant female patients presented for elective C.S for single viable fetus will be included in this study.
* Before anesthesia, the patient will be attached to a monitor of: ECG , heart rate, non invasive blood pressure, pulse taximeter applied on the index finger of the limb not attached to the blood pressure cuff, pulse oximetry and plethysmographic variability index (PVI) and perfusion index (PI) will be taken by (Massimo radical 7, Massimo corp. USA). Measures will be recorded every 5 minutes preoperative.
* Patients with PVI <15 will be excluded from the study.
* Patients with PVI > 15 are started on intravenous infusion of warm ringer lactate solution via suitable pore intravenous cannula to reach target of PVI <15 or a total 1 liter of ringer lactate.
* The patients in which the PVI is corrected by fluid to level below 15 will be Group (C) or corrected group. Patients in which intravenous fluid administration did not result any change in PVI or changed but still higher than 15 will be Group (NC) or non corrected group.

After preoperative preparation patient is shifted to operating theater, with all monitors applied. She will receive spinal block at lumbar 3-4 space with hyperbaric bupivacaine 8 mg plus 25 mic fentanyl. After giving anesthesia and positioning for surgery with a left lateral tilt of 15 degrees,

DETAILED DESCRIPTION:
* This prospective observational study will be carried out on all pregnant women who will undergo elective cesarean section in obstetric department in Tanta university hospitals under spinal anesthesia over four month duration that starts immediately after obtaining ethical committee approval, an informed written consent will be included with the consent for spinal anesthesia for cesarean section, all patients data will be confidential and will be used for the current study only.
* Inclusion criteria:

Pregnant women which are listed to undergo elective caeserian section for single viable baby under spinal anesthesia.

* Exclusion criteria:

  * Patients with pregnancy less than 36 weeks or more than 40 weeks
  * Patients with hypertension , pre-eclampsia , eclampsia.
  * Patients with diabetes
  * Patients with cardiovascular disease and /or arrhythmia.
  * Patients with placenta previa, accreta, percreta.
  * Obese patients with BMI >36
  * Polyhydramnious patients
* On arrival of patients to pre-anaesthesia preparation room, we will allow patients to rest in supine position with 15 degree left tilt by pillow wedge under right hip, after allowing patient to rest for five minutes, measures are recorded: ECG , heart rate, non invasive blood pressure, pulse oximeter applied on the index finger of the limb not attached to the blood pressure cuff, pulse oximetry and Plethysmography variability index (PVI) and perfusion index (PI) will be taken by (Massimo radical 7, Massimo corp. USA). Measures will be recorded every 5 minutes preoperative. Patients with PVI <15 are excluded from the study.

Patients with PVI > 15 are started on intravenous infusion of warm ringer lactate solution via suitable pore intravenous cannula to reach target of PVI <15 or a total 1 liter of ringer lactate.

The patients in which the PVI is corrected by fluid to level below 15 will be Group (C) or corrected group. Patients in which intravenous fluid administration did not result any change in PVI or changed but still higher than 15 will be Group (NC) or non corrected group.

After preoperative preparation patient is shifted to operating theater, with all monitors applied. She will receive spinal block at lumbar 3-4 space with hyperbaric bupivacaine 8 mg plus 25 mic fentanyl. After giving anesthesia and positioning for surgery with a left lateral tilt of 15 degrees, supplemental oxygen at rate of 4 liter/minute is applied.

Measurements will be taken every minute till delivery of the baby, and if the blood pressure is decreased below 20% of the baseline level before anesthesia, patients will be given incremental doses of ephedrine sulfate 0.1 mg /kg till blood pressure normalized above 80% of pre-anesthesia level. All measurements will be recorded in tables and subjected to statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women which are listed to undergo elective caeserian section for single viable baby under spinal anesthesia.

Exclusion Criteria:

* Patients with pregnancy less than 36 weeks or more than 40 weeks, Patients with hypertension , pre-eclampsia , eclampsia, Patients with diabetes, Patients with cardiovascular disease and /or arrhythmia, Patients with placenta previa , accreta, percreta, Obese patients with BMI >36, or Polyhydramnious patients.

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Full term pregnant female patients presented for elective cesarean section delivery of a single viable fetus under spinal anesthesia/
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
The incidence of post-spinal anesthesia hypotension | Through out the whole intraoperative period
  The decrease in the mean arterial pressure below 65 mmHg or below 80% of the baseline value.

SECONDARY OUTCOMES:
The consumption of vasopressors | Through out the whole intraoperative period
  The total dose of ephedrine required to maintain the MAP above 80% of the baseline value

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Ismaiel, M.D, Principal Investigator — Lecturer of Anesthesia and Intensive Care, Tanta University
Locations (2):
- Egypt (2):
  - Tanta University Hospitals, Tanta, Algharbia Governate
  - Tanta University hospitals, Tanta

IPD SHARING:
Plan to Share IPD: Undecided
Once the study had been successfully completed, the data will be shared for other researchers.